CLINICAL TRIAL: NCT04354493
Title: Myoelectric Game Training and Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liberating Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: A-20729; 120180273 (Other: NEIRB)
Record Dates: First submitted 2020-04-17; First posted 2020-04-21 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Amputation; Prosthesis User; Prosthesis
Keywords: myoelectric; training; upper limb; prosthetics; video games

STUDY DESIGN:
Intervention Model Description: Two-group study with same baseline and intervention. One group ceases intervention and returns to control condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Baseline and Training (Experimental): This group consists of a baseline and training conditions only.
  Interventions: Device: Myo-electric Gaming Interface
- Baseline, Training, and Control (Experimental): This group stops training condition sooner and returns to a control to evaluate carry-over effects.
  Interventions: Device: Myo-electric Gaming Interface

INTERVENTIONS:
Device: Myo-electric Gaming Interface — Non-significant risk, video game controller which maps myo-electric control signals to button presses.
  Other Names: MEGI

SUMMARY:
The purpose of this study is to evaluate the effects of myo-electric training tools on prosthesis functional outcomes.

DETAILED DESCRIPTION:
Participants will undergo informed consent and schedule an initial site visit. A logging device will be used to track activity of prosthetic arm usage while in everyday use at home. After a baseline period, participants will schedule a second visit to be introduced to the training technology.

The study will span up to 7 months with participants training at home for 15-60 minutes, 3-5 times a day. Every 3-6 weeks, investigators will schedule a study event and sit visit to conduct functional outcome tasks and measurements.

ELIGIBILITY:
Inclusion Criteria:

* User of upper-limb myo-prosthesis or able to wear prosthesis simulator
* The subjects must be able to read, write, and speak English in order to be properly consented and to express their thoughts to the study personnel, and they must be willing and able to complete the activities outlined in the study.

Exclusion Criteria:

* The risks to pregnant people and fetuses are unknown and therefore pregnant individuals should not participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-04-04 (Actual); Primary Completion 2022-09-18 (Actual); Study Completion 2022-09-18 (Actual)

PRIMARY OUTCOMES:
South Hampton Hand Assesment | 6 week periods
  Hand functional test

SECONDARY OUTCOMES:
Static Tracking Test | 6 week periods
  Myo-electric reach and hold measure.
Dynamic Tracking Test | 6 week periods
  Myo-electric signal path tracing.

CONTACTS AND LOCATIONS:
Locations (1):
- Liberating Technologies Inc., Holliston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided